CLINICAL TRIAL: NCT06094686
Title: Epicardial Adipose Tissue Thickness and the Related Factors in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH5
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; atherosclerosis; epicardial adipose tissue thickness
MeSH Terms: conditions — Spondylitis, Ankylosing; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing spondylitis group: Thirty patients with AS according to the modified New York criteria were included in this cross-sectional study.
  Interventions: Diagnostic Test: epicardial adipose tissue thickness
- Healthy volunteers: Control group was consisted of 31 healthy volunteers
  Interventions: Diagnostic Test: epicardial adipose tissue thickness

INTERVENTIONS:
Diagnostic Test: epicardial adipose tissue thickness — EATT measured via transthoracic echocardiography

SUMMARY:
The aim of this study was to assess the EATT and the related factors in patients with AS and to compare the results with that of the healthy controls'

DETAILED DESCRIPTION:
The aim of this study was to investigate the epicardial adipose tissue thickness (EATT) and the related factors in patients with ankylosing spondylitis (AS) and to compare the results with those of the healthy controls. This cross-sectional study comprised thirty patients diagnosed with AS based on the modified New York criteria. The control group consisted of 31 healthy volunteers. Demographic characteristics were recorded. EATT was measured via transthoracic echocardiography. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Metrology Index (BASMI), Ankylosing Spondylitis Disease Activity Score (ASDAS), Ankylosing Spondylitis Quality of Life (ASQoL), International Physical Activity Questionnaire Short Form (IPAQ-Short Form) were used. Functional capacity assessment was conducted using the six-minute walk test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* Disease duration >1 year,
* Being ≥18 years
* AS diagnosis according to modified New York Criteria

Exclusion Criteria:

* Being illiterate,
* >65 years,
* History of ischemic heart disease,
* Cerebrovascular disease,
* Hypertension,
* Chronic kidney failure,
* endocrinopathies like diabetes mellitus,
* hypothyroidism,
* Cushing syndrome and primary hyperlipidemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with AS that came to Istanbul Physical Medicine and Rehabilitation Education and Research Hospital outpatient clinic between August 2015 and January 2016
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-02 (Actual)

PRIMARY OUTCOMES:
Epicardial adipose tissue thickness | through study completion, an average of 5 months
  Epicardial adipose tissue thickness is measured via transthoracic echocardiography

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index | through study completion, an average of 5 months
  The index indicates that disease activity of AS patients. Higher scores indicate that higher activity
Bath Ankylosing Spondylitis Functional Index | through study completion, an average of 5 months
  The index helps to evaluate disease activity of AS patients. High scores indicate that worse functional status.
Bath Ankylosing Spondylitis Metrology Index | through study completion, an average of 5 months
  The index helps to evaluate spinal mobility of AS patients. Higher scores indicate more limited mobility.
Ankylosing Spondylitis Disease Activity Score | through study completion, an average of 5 months
  This score is used to evaluate disease activity of AS patients. Higher scores indicate that higher activity.
Six minute walk test | through study completion, an average of 5 months
  This test is used to evaluate the patient's functional capacity. In case of low functional capacity, lower scores are observed. Higher scores indicate that higher activity.
Ankylosing Spondylitis Quality of Life | through study completion, an average of 5 months
  it is used for evaluate quality of life of AS patients. A lower score indicates better quality of life
International Physical Activity Questionnaire Short Form | through study completion, an average of 5 months
  it is used for evaluate patient's physical activity. Scoring a high level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Kesiktas, MD, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan to share any data

REFERENCES:
- [Result] Keresztesi AA, Asofie G, Simion MA, Jung H. Correlation between epicardial adipose tissue thickness and the degree of coronary artery atherosclerosis. Turk J Med Sci. 2018 Feb 23;48(1):40-45. doi: 10.3906/sag-1604-58. PMID 29479952
- [Result] Taguchi R, Takasu J, Itani Y, Yamamoto R, Yokoyama K, Watanabe S, Masuda Y. Pericardial fat accumulation in men as a risk factor for coronary artery disease. Atherosclerosis. 2001 Jul;157(1):203-9. doi: 10.1016/s0021-9150(00)00709-7. PMID 11427222
- [Result] Mazurek T, Zhang L, Zalewski A, Mannion JD, Diehl JT, Arafat H, Sarov-Blat L, O'Brien S, Keiper EA, Johnson AG, Martin J, Goldstein BJ, Shi Y. Human epicardial adipose tissue is a source of inflammatory mediators. Circulation. 2003 Nov 18;108(20):2460-6. doi: 10.1161/01.CIR.0000099542.57313.C5. Epub 2003 Oct 27. PMID 14581396